CLINICAL TRIAL: NCT07198698
Title: Effect of Lymphatic Drainage Using the Paloma Sahid Method on Secondary Unilateral Lower Limb Lymphedema in Chilean Adult Women: A Single-Arm Clinical Trial
Brief Title: Sahid Method for Secondary Unilateral Lower Limb Lymphedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDP_SAHID_2025
Record Dates: First submitted 2025-07-18; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema
Keywords: Lymphedema; Manual Lymph Drainage; Lower Extremity
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: A Single-Arm Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental study group (Experimental): Women aged 30 to 65 years diagnosed with lymphedema classified as stage I or II.
  Interventions: Other: Paloma Sahid Method, a patented technique (PCT/CL2023/050061)

INTERVENTIONS:
Other: Paloma Sahid Method, a patented technique (PCT/CL2023/050061) — The participants will receive treatment that integrates manual and mechanical lymphatic drainage through linear sliding movements directed toward relevant lymph nodes. Each session lasts approximately one hour. This intervention was complemented by compression therapy, applying 30-40 mmHg at the ankle, 70% compression at the calf, and 30% compression at the thigh.

SUMMARY:
Manual lymphatic drainage (MLD) is a non-invasive technique frequently used in the management of lymphedema. The Paloma Sahid Method is a patented approach to lymphatic drainage that combines specific manual and mechanical maneuvers and compression. This single-arm clinical trial will evaluate its effects on lower-limb circumference, functional capacity, and quality of life in adult women with secondary unilateral lymphedema.

Thirty-two women aged 30-65 years with stage I-II secondary lymphedema affecting one lower limb will be enrolled through referrals from vascular physicians in public and private centers in the Metropolitan Region of Santiago, Chile. Participants will attend two pre-intervention visits: (1) study information and informed consent; (2) baseline assessments including thermography, body composition and BMI (bioimpedance), blood pressure and heart rate, limb volume by circumferential tape measurements, muscle strength by handheld dynamometry, quality of life (LYMQOL), and function (Lower Extremity Functional Scale, LEFS). A randomized subsample of 10 participants will undergo lymphoscintigraphy before and after treatment to characterize lymphatic circulation.

The intervention consists of 12 sessions of lymphatic drainage using the Paloma Sahid Method, delivered three times per week over one month (about 80 minutes per session). Maneuvers follow linear sliding patterns directed toward regional lymph nodes and are complemented by compression therapy. After completing the 12 sessions, all baseline assessments are repeated.

The primary objective is to determine change in lower-limb circumference from pre- to post-intervention. Secondary objectives include changes in functional capacity, quality of life, thermographic patterns, body composition, muscle strength, hemodynamic measures, and, in the subsample, lymphoscintigraphy findings. The study aims to provide rigorous clinical evidence on a promising, non-surgical option for individuals living with lymphedema.

DETAILED DESCRIPTION:
Background and Rationale Lymphedema involves accumulation of protein-rich interstitial fluid due to impaired lymph transport, commonly leading to limb swelling, tissue changes, recurrent infections, functional limitations, and reduced quality of life. Management is typically multidisciplinary, and non-surgical strategies remain essential. The Paloma Sahid Method (patent code PCT/CL2023/050061) integrates manual and mechanical drainage with standardized linear sliding movements directed toward relevant lymph-node basins, complemented by compression therapy. Despite growing clinical use, robust, prospective evidence on its effects is needed.

Objectives

Primary: Evaluate the effect of lymphatic drainage using the Paloma Sahid Method on lower-limb circumference in adult women with secondary unilateral lymphedema.

Secondary: Assess changes in functional capacity (LEFS), quality of life (LYMQOL), thermographic patterns, body composition and BMI (bioimpedance), muscle strength (handheld dynamometry), resting blood pressure and heart rate, and, in a subsample, lymphoscintigraphy-based lymphatic flow characteristics.

Design and Setting Single-arm clinical trial conducted in Santiago, Chile. Participants attend two pre-intervention visits (consent and baseline testing), receive 12 treatment sessions over ~4 weeks, and complete post-intervention testing.

Participants Women aged 30-65 years with medically diagnosed secondary unilateral lower-limb lymphedema of ≤2 years' duration, classified as stage I or II, able to understand and complete study instruments, and providing informed consent. Key exclusions include inability to complete questionnaires, chronic conditions judged to contraindicate participation (e.g., unstable cardiovascular, pulmonary, autoimmune disease, or diabetes), and absence from more than two consecutive sessions.

Intervention Twelve sessions of lymphatic drainage using the Paloma Sahid Method, delivered three times weekly for one month, approximately 80 minutes per session. The protocol includes manual and mechanical maneuvers with linear sliding toward regional lymph nodes and prescribed compression parameters applied to the limb. Sessions are performed in an outpatient medical center; missed sessions are rescheduled within the same week when possible.

Assessments and Outcomes

Baseline and post-intervention evaluations include:

Anthropometry and composition: BMI and bioimpedance-based body composition.

Hemodynamics: Resting blood pressure and heart rate.

Limb volume: Circumferential tape measurements using a standardized protocol.

Muscle strength: Handheld dynamometry with standardized instructions.

Thermography: Infrared imaging of the lower extremities to describe temperature distribution patterns.

Function and quality of life: LEFS and LYMQOL questionnaires.

Lymphoscintigraphy (subsample, n=10): Pre- and post-intervention imaging to explore lymphatic circulation characteristics.

Primary Outcome Change in lower-limb circumference (affected limb) from pre- to post-intervention.

Secondary Outcomes Changes in LEFS, LYMQOL, thermographic patterns, body composition, muscle strength, blood pressure, heart rate, and lymphoscintigraphy indicators (subsample).

Sample Size and Recruitment A non-probability snowball strategy will be used to recruit 32 women via referrals from peripheral vascular physicians in public and private healthcare centers in the Metropolitan Region. The intervention will be delivered at a medical center located at Avenida La Dehesa 1201, Torre Norte, Office 616, Lo Barnechea.

Statistical Analysis Data will be checked for completeness and plausibility. Normality will be examined (e.g., Shapiro-Wilk). Pre- versus post-intervention changes will be analyzed with Student's t-test or Wilcoxon signed-rank test, as appropriate. Exploratory subgroup analyses (e.g., by age group or lymphedema stage) may be conducted. Two-sided tests and conventional significance levels will be used; effect sizes and confidence intervals will be reported.

Data Management and Quality Assurance Data will be captured in a secure, centralized database with routine backups, anonymization via coded identifiers, and access restricted to authorized personnel. Real-time validation checks will be used to minimize entry errors.

Ethics The protocol was approved by the Interfaculty Scientific Ethics Committee of Universidad Diego Portales on April 16, 2025 (protocol 01-2025). All participants will provide informed consent.

Registration Note Text intentionally omits in-text citations; supporting literature is listed in the References → Citations module of this record.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 30-65 year
* Diagnosed with secondary unilateral lower limb lymphedema less or equal to two years due:surgery, infection, cancer or trauma
* Residing in the Metropolitan Region , Chile
* Having signed informed consent

Exclusion Criteria:

* Inability to understand or respond t questionnaires
* Presence of chronic illnesses such: pulmonary, cardiac, autoimmune disease or diabetes mellitus
* Absence from more than two consecutive sessions

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in lower-limb volume, mL (tape-derived) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Total limb volume (mL) from circumferences every 10 cm (standing). Segmental volume estimated with a truncated-cone approach using adjacent circumferences and 10 cm segment length; total volume is the sum of segments. Higher values indicate greater swelling (worse).

SECONDARY OUTCOMES:
Change in lymphoscintigraphic Transport Index (TI), 0-45 (lower better) | Baseline (within 7 days prior to first session) and Post-intervention (within 7 days after last session)
  Semi-quantitative TI derived from visual criteria on lymphoscintigraphy; range 0-45, with values <10 typical of normal transport; lower scores = better transport. Outcome is pre-post change in TI.
Change in limb temperature difference (ΔT, °C) between affected and contralateral lower limb | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Infrared thermography of predefined regions; ΔT (°C) = affected - contralateral. Positive values indicate higher temperature on the affected limb. Outcome is change in ΔT.
Change in Lower Extremity Functional Scale (LEFS) total score, 0-80 (higher better) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  LEFS: 20 items scored 0-4; total 0-80; higher scores indicate better function. Outcome is change in total score.
Change in knee extensor isometric strength, kg | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Handheld dynamometry in standardized position; three trials, maximum value (kg) retained. Outcome is change in kg.
Change in Fagerström Test for Nicotine Dependence (FTND) total score, 0-10 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  FTND total score 0-10; higher scores indicate greater nicotine dependence. Outcome is change in total score.
Mean resting systolic blood pressure during the intervention, mmHg | During the 4-week intervention (12 sessions)
  Measured each session after ≥5 min seated rest; two readings averaged per session. Outcome is the per-participant mean (mmHg) across 12 sessions.
Mean resting diastolic blood pressure during the intervention, mmHg | During the 4-week intervention (12 sessions)
  Measured each session after ≥5 min seated rest; two readings averaged per session. Outcome is the per-participant mean (mmHg) across 12 sessions.
Mean resting heart rate during the intervention, bpm | During the 4-week intervention (12 sessions)
  Measured each session after ≥5 min seated rest; outcome is the per-participant mean (bpm) across 12 sessions.
Change in Lymphedema Quality of Life (LYMQOL)-Leg Symptoms domain score, 1-4 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  LYMQOL-Leg domain mean score; 1-4; higher = worse. Outcome is change in domain score.
Change in Lymphedema Quality of Life (LYMQOL)-Leg Function domain score, 1-4 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Domain mean; higher = worse. Outcome is change in domain score.
Change in Lymphedema Quality of Life (LYMQOL)-Leg Appearance domain score, 1-4 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Domain mean; higher = worse. Outcome is change in domain score.
Change in Lymphedema Quality of Life (LYMQOL)-Leg Emotion domain score, 1-4 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Domain mean; higher = worse. Outcome is change in domain score.
Change in Lymphedema Quality of Life (LYMQOL)-Leg overall quality of life, Visual Analog Scale (VAS), 0-10 (higher better) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Self-rated overall QoL on 0-10 VAS; higher = better. Outcome is change in VAS.
Change in body mass index (BMI), kg/m² | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  BMI = weight/height² (kg/m²). Outcome is change in BMI.
Change in body fat percentage, % | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Bioelectrical impedance under standardized pretest conditions. Outcome is change in % body fat.
Change in skeletal muscle mass, kg | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Derived from bioelectrical impedance; outcome is change in kg.
Change in body weight, kg | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  Calibrated digital scale; outcome is change in kg.
Standing height, cm (baseline only) | Baseline (within 7 days prior to first session)
  Stadiometer; height recorded in cm at baseline for BMI calculation.
Change in pain intensity, Visual Analog Scale (VAS), 0-10 (higher worse) | Baseline (within 7 days prior to first session) and Week 4 (within 7 days after last session)
  10-cm VAS anchored at 0 = no pain and 10 = worst imaginable; outcome is change in score.
Participants with intervention-related adverse events | From first intervention session through Week 4 (study completion)
  Number of participants reporting events plausibly related to treatment (e.g., musculoskeletal discomfort, dizziness, falls), recorded during sessions and between-session reports.

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Sahid, Bachelor, Principal Investigator — University Diego Portales
Locations (1):
- Av. La Dehesa 1201, Torre Norte, Of. 616, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The cohort is small and potentially re-identifiable, and the informed consent and ethics approval (UDP CEI 01-2025) do not authorize external sharing of individual-level data. Aggregate results will be reported. Study documents (e.g., protocol, analysis code, data dictionary) may be provided upon request.

REFERENCES:
- [Background] Young SS, Schilling AM, Skeans S, Ritacco G. Short duration anaesthesia with medetomidine and ketamine in cynomolgus monkeys. Lab Anim. 1999 Apr;33(2):162-8. doi: 10.1258/002367799780578363. PMID 10780820
- [Background] Yue H, Devidas S, Guggino WB. The two halves of CFTR form a dual-pore ion channel. J Biol Chem. 2000 Apr 7;275(14):10030-4. doi: 10.1074/jbc.275.14.10030. PMID 10744680
- [Background] Kincaid HL Jr, Jirgensons B. Circular dichroism of kappa- and lambda type Bence-Jones proteins at various pH values and temperatures. Biochim Biophys Acta. 1972 Jun 22;271(1):23-33. doi: 10.1016/0005-2795(72)90129-8. No abstract available. PMID 4624940
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Hwang JH, Choi JY, Lee JY, Hyun SH, Choi Y, Choe YS, Lee KH, Kim BT. Lymphscintigraphy predicts response to complex physical therapy in patients with early stage extremity lymphedema. Lymphology. 2007 Dec;40(4):172-6. PMID 18365531
- [Background] International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2013 Consensus Document of the International Society of Lymphology. Lymphology. 2013 Mar;46(1):1-11. PMID 23930436
- [Background] Yamamoto T, Matsuda N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. The earliest finding of indocyanine green lymphography in asymptomatic limbs of lower extremity lymphedema patients secondary to cancer treatment: the modified dermal backflow stage and concept of subclinical lymphedema. Plast Reconstr Surg. 2011 Oct;128(4):314e-321e. doi: 10.1097/PRS.0b013e3182268da8. PMID 21921744
- [Background] Arrive L, Derhy S, El Mouhadi S, Monnier-Cholley L, Menu Y, Becker C. Noncontrast Magnetic Resonance Lymphography. J Reconstr Microsurg. 2016 Jan;32(1):80-6. doi: 10.1055/s-0035-1549133. Epub 2015 Mar 31. PMID 25826439
- [Background] Cormier JN, Askew RL, Mungovan KS, Xing Y, Ross MI, Armer JM. Lymphedema beyond breast cancer: a systematic review and meta-analysis of cancer-related secondary lymphedema. Cancer. 2010 Nov 15;116(22):5138-49. doi: 10.1002/cncr.25458. PMID 20665892
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Thomas C, Le JT, Benson E. Managing Lymphedema in Fracture Care: Current Concepts and Treatment Principles. J Am Acad Orthop Surg. 2020 Sep 15;28(18):737-741. doi: 10.5435/JAAOS-D-19-00722. PMID 32618680
- [Background] Basta MN, Gao LL, Wu LC. Operative treatment of peripheral lymphedema: a systematic meta-analysis of the efficacy and safety of lymphovenous microsurgery and tissue transplantation. Plast Reconstr Surg. 2014 Apr;133(4):905-913. doi: 10.1097/PRS.0000000000000010. PMID 24352208
- See also: Pereira N.,Venegas J. y Cifuentes I. Calidad de Vida en pacientes sometidos al tratamiento quirúrgico del linfedema. Validación lingüística y adaptación transcultural del Lymphedema Quality of Life Score (LeQOLiS). Rev. cir. 2020, vol. 72, n. 2, pp. 113- — https://www.revistacirugia.cl/index.php/revistacirugia/article/view/465
- See also: Orientación Técnica Programa de Salud Cardiovascular 2017.Criterios programa salud cardiovascular. ANEXO 5. Perfil de presión arterial. Técnica estandarizada de medición automática de la presión arterial. — https://capacitacionesonline.com/wp-content/uploads/2017/09/Programa-de-salud-cardiovascular.-MINSAL-Chile-2017.pdf